CLINICAL TRIAL: NCT05352152
Title: Application of Next Generation Sequence in the Etiological Diagnosis of Abdominal Infection in Patients With Liver Disease
Brief Title: Application of NGS in Ascites Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Zhangdz2022
Record Dates: First submitted 2022-04-23; First posted 2022-04-28 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Ascites Infection; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ascites infection: Patients who is confirmed with ascites infection or clinically diagnosed as ascites infection will be enrolled in this cohort.
  Interventions: Diagnostic Test: Next generation sequence

INTERVENTIONS:
Diagnostic Test: Next generation sequence — Next generation sequence will be used to detect the pathogens in ascites.
  Other Names: Traditional detection method

SUMMARY:
Liver cirrhosis is a common serious chronic disease. There are about 123 million patients with liver cirrhosis worldwide, and about 1 million people die of liver cirrhosis every year. The proportion of bacterial infection in hospitalized patients with liver cirrhosis is between 25% and 46%, among which spontaneous bacterial peritonitis (SBP) is the most common type of infection in patients with liver cirrhosis. After early and reasonable diagnosis and treatment, the mortality of cirrhotic patients with SBP can be reduced from more than 90% to about 20%. Therefore, rapid and accurate diagnosis is of great help to improve the prognosis of cirrhotic patients with SBP. However, at present, the traditional detection methods is time-consuming with a low detection rate, and can not detect intracellular bacteria and some other types of pathogens.

Next-generation sequencing (NGS) is a relatively new detection technology which can detect the nucleic acid sequence information in a high-throughput, large-scale way. It can detect the pathogens comprehensively, fast and accurately. In recent years, NGS has gradually transitioned from a research tool to a diagnostic method. Many studies have shown that NGS has better application value in bloodstream infections, ocular infectious diseases, central nervous system infectious diseases and respiratory infectious diseases. However, there is still a lack of research on the use of NGS for the detection of pathogenic microorganisms in ascites. Therefore, by comparing the next generation sequence (NGS) and traditional detection technology in the detection of pathogens in ascites, this study aimed to evaluate the value of NGS in the pathogenic diagnosis of ascites infection.

DETAILED DESCRIPTION:
This study is observational and approximately 50 subjects will be included according to inclusion and exclusion criteria. Patients who meet the inclusion and exclusion criteria, will be were collected a sufficient amount of ascites, and the collected ascites will be divided into four different groups. One group will be used as a control, and the other three groups will be centrifugated at different speeds. After centrifugation, the four groups of specimens will be tested by NGS to detect the pathogens. By comparing the detection rate of NGS test for concentrated samples and unconcentrated samples, and this study aims to observe whether centrifugation could increase the detection rate. By comparing the results of NGS and the results of traditional detection methods, this study also aims to explore the consistency between NGS and traditional detection methods, and whether NGS has higher detection rates.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign informed consent;
2. Age ≥ 18 years old;
3. Have full civil capacity;
4. The amount of ascites is suitable for puncture;
5. Ascites infection confirmed by clinical etiology test or clinically suspected ascites infection (such as elevated leukocyte count, elevated procalcitonin, abdominal inflammation indicated by imaging, etc.)

Exclusion Criteria:

1. Those who cannot cooperate with the test;
2. Those whose samples cannot be obtained by puncture;
3. The cause of ascites is clear;
4. Those who are considered to be not suitable for this study

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ascites infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-04-25 (Estimated)

PRIMARY OUTCOMES:
Results of next generation sequence | within 10 days of patient enrollment in study
  Pathogens detected by NGS
Results of traditional detection methods | within 10 days of patient enrollment in study
  Pathogens detected by traditional detection methods

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Zhang, M.D., Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No